CLINICAL TRIAL: NCT02511093
Title: A Team-Based Care for Hypertension Management (TBC-HTA): A Randomized Controlled Study
Brief Title: A Team-Based Care for Hypertension Management (TBC-HTA)
Acronym: TBC-HTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other); Université du Québec à Trois-Rivières (Other); McGill University (Other)
Responsible Party: Principal Investigator, Valérie Santschi, Dr. Valérie Santschi, PharmDipl, PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 449/13
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
Keywords: Hypertension; Team-based care; Collaboration; Healthcare professionals; Healthcare services
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBC intervention (Experimental): A structured collaborative intervention delivered by trained nurses of ambulatory clinics and by community pharmacists working in collaboration with physicians during 6-month of follow-up includes:
  * BP measurements;
  * an educational and counselling intervention on patient adherence;
  * an educational and counselling intervention on lifestyle (physical activity and diet).
  Physicians adjust antihypertensive medications based on nurse and pharmacist feedback.
  Interventions: Behavioral: TBC intervention
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: TBC intervention — A structured collaborative intervention delivered by trained nurses of ambulatory clinics and by community pharmacists working in collaboration with physicians during 6-month of follow-up includes:
  * BP measurements;
  * an educational and counselling intervention on patient adherence;
  * an educational and counselling intervention on lifestyle (physical activity and diet) Physicians adjust antihypertensive medications based on nurse and pharmacist feedback.
  Arms: TBC intervention

SUMMARY:
The purpose of this study is to determine whether a team-based care (TBC) intervention, combining physician, nurse and pharmacist care improves BP control compared to usual care at 6 months among outpatients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* treated patients with uncontrolled hypertension (defined as daytime systolic/diastolic ambulatory blood pressure monitoring (ABPM) ≥135/85mmHg) taking one or two antihypertensive medications;
* speak and understand French;
* agree to use the same pharmacy's services for the whole duration of the study.

Exclusion Criteria:

* unable to understand the study aim;
* pregnancy and lactating;
* livimg in a nursing home;
* hospitalization during the recruitment period;
* participation in another study;
* daytime ABPM>180/110 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Difference in daytime ABPM at 6-month between TBC and usual care patients | 6-month
  Difference in daytime ABPM at 6-month between TBC and usual care patients
Difference in the proportion of patients with controlled blood pressure (daytime ABPM <135/85 mmHg) at 6-month between TBC and usual care patients | 6-month
  Difference in the proportion of patients with controlled blood pressure (daytime ABPM <135/85 mmHg) at 6-month between TBC and usual care patients

SECONDARY OUTCOMES:
Patients and healthcare professionals' acceptance and satisfaction with the TBC-intervention | 6-month
  Patients and healthcare professionals' acceptance and satisfaction with the TBC-intervention
Difference in the proportion of TBC and usual care patients with controlled blood pressure (daytime ABPM <135/85 mmHg) at 12-month (6 months after intervention stopped) | 12-month
  Difference in the proportion of TBC and usual care patients with controlled blood pressure (daytime ABPM <135/85 mmHg) at 12-month (6 months after intervention stopped)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Santschi, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Michel Burnier, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Service de Néphrologie et Hypertension, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Santschi V, Wuerzner G, Pais B, Chiolero A, Schaller P, Cloutier L, Paradis G, Burnier M. Team-Based Care for Improving Hypertension Management: A Pragmatic Randomized Controlled Trial. Front Cardiovasc Med. 2021 Oct 25;8:760662. doi: 10.3389/fcvm.2021.760662. eCollection 2021. PMID 34760950
- [Derived] Santschi V, Wuerzner G, Chiolero A, Burnand B, Schaller P, Cloutier L, Paradis G, Burnier M. Team-based care for improving hypertension management among outpatients (TBC-HTA): study protocol for a pragmatic randomized controlled trial. BMC Cardiovasc Disord. 2017 Jan 21;17(1):39. doi: 10.1186/s12872-017-0472-y. PMID 28109266